CLINICAL TRIAL: NCT03017846
Title: Safety and Efficacy of Topical Cantharidin for the Treatment of Molluscum Contagiosum, Phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven R Cohen (Other)
Responsible Party: Sponsor-Investigator, Steven R Cohen, Professor, Montefiore Medical Center
Organization: Montefiore Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-10-195
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — Cantharidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cantharidin Treatment (Experimental): Subjects with lesions treated with topical cantharidin every 3 weeks up to 12 weeks.
  Interventions: Drug: Cantharidin

INTERVENTIONS:
Drug: Cantharidin — Application of topical cantharidin

SUMMARY:
Cantharidin is cited in the dermatology and pediatric literature as a valuable treatment option. Treatment is often available in private practice offices, where a prescribing physician may offer a non-FDA approved treatment on an individualized basis. The situation is different in many hospital and academic settings, such as our own for example, where the formulary is defined through a FDA-approved indication. The absence of an indication precludes its addition to many hospital formularies, thus limiting the options available to a prescribing physician and denying patient access to a treatment offered in the private practice setting. An indication and formulary status require controlled clinical trials on the safety and efficacy of cantharidin in MC. The objective of this trial is to see if this commercially-viable cantharidin formulation has a comparable safety and efficacy profile as formulations previously studied under conditions which most closely match the what has been historically done in the clinic.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of MC by the Principal Investigator.

Maximum of 50 lesions on locations including the face, trunk, back, left or right arm, left or right leg, hands, feet, buttocks, and groin.

Execution of Informed Consent and or assent forms

Exclusion Criteria:

Patients with immunosuppression, including organ transplantation, HIV infection.

Patients utilizing immunosuppressive agents (including oral corticosteroids) will be excluded except for patients using inhaled corticosteroids, such as those utilized for asthma or allergic rhinitis.

Females who have reached menarche and are sexually active as well as pregnant patients will be excluded as the effects of this drug have not been evaluated in pregnancy.

Patients who have greater than 50 MC lesions will also be excluded from the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Cohen, MD, MPH, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cantharidin Treatment
Started | 30
Completed | 25
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cantharidin Treatment
Number analyzed (Participants) | 30
Age, Customized [Count of Participants; unit: Participants]
  Age 1-3 years | 6
  Age 4-6 years | 11
  Age 7-10 years | 12
  Age 11-13 years | 1
  Age 14-17 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0
  Asian | 0
  Caucasian | 3
  Hispanic | 17
  Other | 9
  Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Lesion Clearance
Description: 100% reduction in baseline lesion count
Time Frame: Assessed at each visit, until final visit on week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cantharidin Treatment
Number analyzed (Participants) | 30
Participants | 11

2. Secondary Outcome: Number of Subjects Who Achieve a Clearance of at Least 90% of Their Molluscum Lesions
Time Frame: At study completion, up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cantharidin Treatment
Number analyzed (Participants) | 27
Participants | 14

3. Secondary Outcome: Change in the Total Children's Dermatology Life Quality Index Score
Description: Change in the Total Children's Dermatology Life Quality Index (CDLQI) given Visit 1 prior to the first treatment and at the last study visit, up to 12 weeks. The CDLQI examines how the patient feels about the symptoms and treatment, as well as how it affects leisure, school, personal relationships, sleep, clothing choices. A total score is calculated.
  The total score for the CDLQI scores range:
  0-1 = no effect on child's life 2-6 = small effect 7-12 = moderate effect 13-18 = very large effect 19-30 = extremely large effect
Time Frame: Baseline (At beginning of study, before treatment) and end of study (at study completion, week 12 or at earlier visit if all lesions have cleared)
Population: All patients who were not lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cantharidin Treatment
Number analyzed (Participants) | 27
score on a scale
  At beginning of study, before treatment | 3.9 (5.6)
  At end of study | 0.38 (1.3)

4. Secondary Outcome: Number of Patients Achieving Complete Lesion Clearance Compared to Prior Study (NCT02665260)
Description: Comparison of the number of subjects achieving complete lesion clearance at study completion (up to 12 weeks) to the same measure obtained in our previous study (NCT02665260)
Time Frame: At study completion, up to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Current Study: Subjects with lesions treated with topical cantharidin every 3 weeks up to 12 weeks in the present study.
  Cantharidin: Application of topical cantharidin
- NCT02665260: Subjects with lesions treated with topical cantharidin every 3 weeks up to 12 weeks in the previous study NCT02665260.
  Cantharidin: Application of topical cantharidin
Arm/Group | Current Study | NCT02665260
Number analyzed (Participants) | 25 | 23
Participants | 11 | 7

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, up to 12 weeks.
Arm/Group | Cantharidin Treatment
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 28/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cantharidin Treatment (N=30)
Constipation (Gastrointestinal disorders) | 1 (1)
Tooth Fracture (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Application Site Discoloration (Skin and subcutaneous tissue disorders) | 12 (12)
Application Site Vesicles (Skin and subcutaneous tissue disorders) | 21 (21)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6)
Excoriation (Skin and subcutaneous tissue disorders) | 2 (2)
Impetigo (Skin and subcutaneous tissue disorders) | 1 (1)
Skin pain (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03017846/Prot_SAP_000.pdf